CLINICAL TRIAL: NCT01750840
Title: A Clinical Registry to Collect Patient Outcome Data for the BIOMET® EBI Bone Healing System, BIOMET® OrthoPak® Non-invasive Bone Growth Stimulator System, and the BIOMET® SpinalPak® Non-Invasive Spine Fusion Stimulator System
Brief Title: A Clinical Registry to Collect Patient Outcome Date for the BIOMET® Stimulator Systems
Status: Terminated | Type: Observational
Why Stopped: Slow enrollment and poor patient follow-up following enrollment
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CS-101P
Record Dates: First submitted 2012-12-13; First posted 2012-12-17 (Estimated); Results first posted 2016-06-14 (Estimated); Last update posted 2017-06-19 (Actual); Status verified 2017-06

CONDITIONS: Fusion of Spine (Disease); Fractures, Ununited
MeSH Terms: conditions — Disease; Fractures, Ununited

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Stimulation Group: All patients will receive either the Biomet® EBI Bone Healing System, Biomet OrthoPak® Non-invasive Bone Growth Stimulator System or Biomet SpinalPak® Non-Invasive Spine Fusion Stimulator Systems.
  Interventions: Device: Biomet® EBI Bone Healing System; Device: Biomet Orthopak® Non-Invasive Bone Growth Stimulator System; Device: Biomet SpinalPak® Non-Invasive Spine Fusion Stimulator

INTERVENTIONS:
Device: Biomet® EBI Bone Healing System — A pulsed electromagnetic fields electrical stimulation device used for the treatment of fracture nonunions. Designed to be used for 3-10 hours per day with a recommended use of 10 hours per day.
Device: Biomet Orthopak® Non-Invasive Bone Growth Stimulator System — A capacitive coupling electrical stimulation device used for the treatment of fracture nonunions. Designed to be used for 24 hours per day.
Device: Biomet SpinalPak® Non-Invasive Spine Fusion Stimulator — A capacitive coupling electrical stimulation device used as an adjunctive treatment to lumbar spinal fusion. Designed to be used for 24 hours per day.

SUMMARY:
The purpose of this clinical registry is to capture data on an ongoing basis from a population of patients who will use Biomet's BHS, OrthoPak and SpinalPak devices.

DETAILED DESCRIPTION:
The purpose of this clinical registry is to capture current, real-world, bone specific healing data from the medical records of patients being treated with a Biomet® EBI Bone Healing System (BHS), the Biomet® OrthoPak® Non-Invasive Bone Growth Stimulator System, or the Biomet® SpinalPak® Non-Invasive Spine Fusion Stimulator System. This study will provide current data on the effectiveness of these electrical stimulation devices.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has agreed to undergo electrical stimulation therapy as prescribed by their physician.
2. Subject has agreed to return to the physician for their physician required follow up visits.
3. Subject will undergo treatment with Biomet's BHS, OrthoPak or SpinalPak devices.
4. Subject has agreed to complete QoL questionnaires prior to starting treatment and at the follow up visit when the physician has determined the subject to be either healed or failed.

Exclusion Criteria:

1. Any subject not willing to comply with the physician prescribed treatment program and follow up visit schedule.
2. Any subject not willing to complete the QoL questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This clinical registry will be a prospective, multi-center study. Subjects will undergo treatment with Biomet's BHS or OrthoPak devices for non-spinal applications.
  Subjects will undergo treatment with Biomet's SpinalPak for spinal applications
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2012-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randy Graham, Study Director — Zimmer Biomet
Locations (1):
- Cumberland Orthopedics, Vineland, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Stimulation Group: All patients will receive either the Biomet EBI Bone Healing System, Biomet OrthoPak Non-invasive Bone Growth Stimulator System or Biomet SpinalPak Non-Invasive Spine Fusion Stimulator Systems.
Period: Overall Study
Arm/Group | Stimulation Group
Started | 8
Completed | 4
Not Completed | 4
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Arm/Group | Stimulation Group
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 40 [9 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Assessment of Healing
Description: Bone healing was assessed on x-rays and/or CT scan.
Time Frame: The time frame for healing determination was not pre-specified. Patients were evaluated at regular doctors' visits for up to 12 months. The physician determined the time point at which healing occurred for each patient at their regular visits.
Population: All patients, with one nonunion fracture each, were treated with the Biomet EBI Bone Healing System. Four patients had final healing outcomes reported (two patients with a 5th metatarsal nonunion, one patient with a tibial nonunion and one patient with a fibula nonunion) and all healed in an average time of 2.5 months.
Measure: Number; unit: percentage of healed fractures
Units Other Than Participants: Fractures
Arm/Group | Stimulation Group
Number analyzed (Participants) | 4
Number analyzed (Fractures) | 4
percentage of healed fractures | 100

2. Secondary Outcome: Quality of Life Assessment
Description: Quality of life was intended to be measured by 5 scoring systems that ask a range of questions about the patient's pain and function. No quality of life data was captured for any of the patients and as such no quality of life analysis was performed.
Time Frame: The quality of life assessment was to be completed at the regular doctor's visit at which the physician determined the patient to be healed. No quality of life data was collected.
Population: No quality of life data was collected for any of the patients enrolled in the study. As such, no analysis was performed on quality of life measures.
Groups:
- Stimulation Group: All patients will receive either the Biomet EBI Bone Healing System, Biomet OrthoPak Non-invasive Bone Growth Stimulator System or Biomet SpinalPak Non-Invasive Spine Fusion Stimulator Systems.
  Biomet EBI Bone Healing System: A pulsed electromagnetic fields electrical stimulation device used for the treatment of fracture nonunions. Designed to be used for 3-10 hours per day with a recommended use of 10 hours per day.
  Biomet Orthopak Non-Invasive Bone Growth Stimulator: A capacitive coupling electrical stimulation device used for the treatment of fracture nonunions. Designed to be used for 24 hours per day.
  Biomet SpinalPak Non-Invasive Spine Fusion Stimulator System: A capacitive coupling electrical stimulation device used as an adjunctive treatment to lumbar spinal fusion. Designed to be used for 24 hours per day.
Arm/Group | Stimulation Group
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the entire period that each of the patients was followed. Patients were followed up to 1 year.
Arm/Group | Stimulation Group
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No